CLINICAL TRIAL: NCT05109715
Title: The Effect of Mechanical Ventilation on the Occurrence of Myocardial Ischemia in Patients Undergoing Endoscopic Coronary Artery Bypass Grafting (Endo-CABG): a Pilot Study
Brief Title: The Effect of Mechanical Ventilation on the Occurrence of Myocardial Ischemia: a Pilot Study
Acronym: VENTMICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: f/2021/118
Record Dates: First submitted 2021-10-27; First posted 2021-11-05 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Myocardial Ischemia; Hypoxia
Keywords: Cardiac surgery; Ventilation
MeSH Terms: conditions — Myocardial Ischemia; Hypoxia; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Ventilation is discontinued after going on CPB and lungs are exposed to atmospheric pressure.
  Blood will be drawn:
  * At baseline: before general anaesthesia
  * After start of heart-lung machine
  * After clamping the aorta
  * Before unclamping the aorta
  * After the operation
  * 5 h after clamping the aorta
  * 12 hours after clamping the aorta
  * 24 hours after aortic clamping
  * 48h after clamping the aorta
  * 72 hours after clamping the aorta
  Interventions: Procedure: Discontinued ventilation
- Ventilation group (Experimental): Ventilation is continued from going on CPB until clamping of the ascending aorta.
  Blood will be drawn:
  * At baseline: before general anaesthesia
  * After start of heart-lung machine
  * After clamping the aorta
  * Before unclamping the aorta
  * After the operation
  * 5 h after clamping the aorta
  * 12 hours after clamping the aorta
  * 24 hours after aortic clamping
  * 48h after clamping the aorta
  * 72 hours after clamping the aorta
  Interventions: Procedure: Continued ventilation

INTERVENTIONS:
Procedure: Continued ventilation — Ventilation is continued from going on CPB until clamping of the ascending aorta with tidal volume 3ml/kg ideal body weight, Fraction of inspired oxygen (FiO2) 50%, respiratory rate 5/min and Inspiratory:Expiratory (I/E) ratio 1/2.
  Arms: Ventilation group
Procedure: Discontinued ventilation — Ventilation is discontinued after going on CPB and lungs are exposed to atmospheric pressure
  Arms: Control group

SUMMARY:
The goal of the proposed pilot study is to determine which method can detect myocardial ischemia at the predefined timepoints during endo-CABG. Additionally, the investigators want to examine the influence of mechanical ventilation on the occurrence of myocardial ischemia in patients undergoing endo-CABG.

DETAILED DESCRIPTION:
CABG is the most effective therapy for patients suffering from coronary artery disease, a condition which annually affects 126 million people worldwide. During this surgery, cardiopulmonary bypass (CPB) takes over the function of the heart and lungs. As a result of the emergence of minimally invasive cardiac surgery (MICS) (e.g. endoscopic-CABG), peripheral CPB with femoral arterial cannulation became the most commonly utilized strategy. However, the use of retrograde arterial perfusion is not without risk. It may result in the upper body and coronary arteries being perfused with deoxygenated blood. The hypoxemia will induce myocardial ischemia and this can harm the cardiac myocytes. A solution for this inconvenience is still lacking. Literature reports that establishing adequate ventilation support should help overcome this phenomenon. However, this approach has not yet been investigated in a clinical trial. In general, this phenomenon is not well recognized in the typical surgical setting, and limited research has been done.

The goal of the proposed pilot study is to determine which method can detect myocardial ischemia at the predefined timepoints during endo-CABG. Additionally, the investigators want to examine the influence of mechanical ventilation on the occurrence of myocardial ischemia in patients undergoing endo-CABG.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patients undergoing their first elective endo-CABG procedure
* Patients capable of signing the informed consent
* Patients able to speak Dutch or French

Exclusion Criteria:

* Ongoing participation in another trial
* Ejection fraction < 50%
* Lung diseases (COPD, asthma)
* Use of corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
The detection of myocardial ischemia using Cardiac Troponin T (cTn-T) | Until 72 hours after clamping the aorta
  If the value of Cardiac Troponin T (cTn-T) exceeds 14 ng/L, then cTn-T is able to detect myocardial ischemia at the predefined time points.
The detection of myocardial ischemia using Heart-type Fatty Acid Binding Protein (hFABP) | Until 5 hours after clamping the aorta
  If the value of Heart-type Fatty Acid Binding Protein (hFABP) exceeds 6 ng/L, then hFABP is able to detect myocardial ischemia at the predefined time points.
The detection of myocardial ischemia using Creatine Kinase Myocardial Band (CK-MB) | Until 48 hours after clamping the aorta
  If the value of Creatine Kinase Myocardial Band (CK-MB) exceeds 6.2 µg/L, then CK-MB is able to detect myocardial ischemia at the predefined time points.
The detection of myocardial ischemia using Reactive Oxygen Species (ROS) | Until unclamping the aorta (on average until 64 minutes after clamping the aorta)
  Reactive Oxygen Species (ROS) measurements include a malondialdehyde assay to assess the lipid peroxidation, an Oxystat test to analyse the total peroxide levels and a protein carbonyl assay to assess the protein damage due to cardiomyocyte dysfunction. Additionally a biopsy will be taken to analyze pro- and anti-oxidants. If a significant increase in lipid peroxidation, total peroxide levels, protein damage and/or pro- and anti-oxidants in the ventilation group compared to the control group is present, then ROS is able to detect myocardial ischemia at the predefined time points.
The occurence of hypoxemia using blood gas measurement | Until the end of surgery (on average until 203 minutes after the start of the surgery)
  If the partial pressure of oxygen (PaO2) is lower than 60 mmHg, then hypoxemia is present.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Kaya, PhD, Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No